CLINICAL TRIAL: NCT01446549
Title: Quantitative Modeling of Motor Performance in Parkinson's Disease After High Intensive Antigravity Locomotor Exercise or Deep Brain Stimulation
Brief Title: Motor Performance in Parkinson's Disease After High Intensive Exercise or Deep Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other); Bispebjerg Hospital (Other); Danish Parkinson Association (Other)
Responsible Party: Principal Investigator, Martin Hoyer Rose, Principal Investigator, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2010-051
Record Dates: First submitted 2011-09-29; First posted 2011-10-05 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Experimental)
  Interventions: Procedure: Deep Brain Stimulation
- Locomotor Exercise (Experimental)
  Interventions: Other: High intensive antigravity locomotor exercise

INTERVENTIONS:
Other: High intensive antigravity locomotor exercise — High intensive antigravity locomotor exercise, 3 sessions/week, for 8 weeks.
  Arms: Locomotor Exercise
Procedure: Deep Brain Stimulation — Deep Brain Stimulation implantation
  Arms: Deep Brain Stimulation

SUMMARY:
The purpose of this study is (1) to provide quantitative information of the motor manifestations of Parkinson's disease and (2) to quantify the effect of high intensive antigravity locomotor exercise or Deep Brain Stimulation implantations in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria (exercise arm):

* Idiopathic Parkinson's disease
* A stable condition the last 6 months
* Hoehn and Yahr 2 - 3

Inclusion Criteria (Deep Brain Stimulation arm):

* Patients referred to Deep Brain Stimulation

Exclusion Criteria:

* Cardiovascular disease
* Conditions that contraindicate physical exercise or the examination

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in Isometric Tremor Approximate Entropy | Change from baseline up to 16 weeks
  Approximate Entropy is a metric. When used to quantify isometric tremor irregularity, information of dominant/pathological CNS oscillators can be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Rose, MSci, Principal Investigator — Department of Exercise and Sport Sciences, University of Copenhagen; Bente R Jensen, MSci, PhD, Study Chair — Department of Exercise and Sport Sciences, University of Copenhagen; Stig Sonne-Holm, MD, DSc, Study Chair — Department of Orthopedic Surgery, Hvidovre University Hospital; Annemette Løkkegaard, MD, PhD, Study Chair — Department of Neurology, Bispebjerg University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark